CLINICAL TRIAL: NCT01953458
Title: Therapeutic Option for Hepatitis B and C: a French Cohort
Acronym: HEPATHER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Bristol-Myers Squibb (Industry); Gilead Sciences (Industry); Janssen-Cilag Ltd. (Industry); Merck Sharp & Dohme LLC (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: ANRS CO22 HEPATHER; 2011-A01438-33 (Other: ID RCB)
Record Dates: First submitted 2013-09-19; First posted 2013-10-01 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Viral Hepatitis B; Viral Hepatitis C
Keywords: Hepatitis B and C; ANRS HEPATHER French Cohort
MeSH Terms: conditions — Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- hepatitis C and/or B

SUMMARY:
* The cohort will integrate clinical, genetic, pharmacogenomics, environmental, biomarkers and behavioral data in a large number of patients and will be a leading equipment for crossdisciplinary and translational research on hepatitis.
* The cohort will be the main support for estimating the relative effects of treatments and for further cost-effectiveness studies on the management and treatment options in chronic HCV (Hepatitis C Virus)and HBV (Hepatitis B virus)infections.

DETAILED DESCRIPTION:
General schedule of the study :

* Prospective multicenter national study
* Duration of inclusions:3 years
* Effective : 25000 patients
* Duration of the follow-up: 7-8 years
* Duration of the cohort: 10 years

Population :

Twenty-five thousands of people will be included and followed in investigator sites, 15000 with an hepatitis C and 10000 with an hepatitis B, according their usual follow-up of their liver disease.

We aim to include up to 50% patients naive of any HCV treatment at inclusion. Also HBV "cured" patients could be included (less than 10%).

Design study:

* During the recruitment visit, demographics, clinical, biological and virological data will be collected. The patient will move through several assessments involving questionnaires, measurements and blood sampling.
* Then the minimum follow-up is one medical visit per year. The follow-up (clinical data and biological collections) will be driven by events or based on protocols that will be developed on the cohort.
* There is no specific treatment in this cohort.

The scientific project is structured into 4 scientific thematic axes :

* Therapeutics:

  * To analyze the long term effects of therapy
  * To study predictors of virological response or fibrosis progression (or regression)and pharmacokinetic/pharmacodynamics either in HCV or HBV treatments
* Virology:

  * To understand the molecular mechanisms of antiviral treatment success and failure
  * To provide treatment recommendation to prevent resistance and achieve sustained or definitive control of infection
* Pathology and physiopathology :

  * To identify new pathophysiological targets responsible for chronic hepatitis severity,prognosis, and evolution.
  * To validate new therapeutic combinations based on pathophysiological researches
* Public Health:

  * To identify psychosocial and behavioral correlates of access to care, progression of liver disease and of the burden of chronic viral hepatitis B and C.
  * To evaluate the cost-effectiveness of HBV and HCV treatments and quality of life

ELIGIBILITY:
Inclusion Criteria:

* HBV-positive patients

  * Chronic hepatitis B defined by a positive HBsAg ( surface antigen of the hepatitis B virus) for at least 6 months
  * Acute hepatitis B defined as a recent appearance (<6 months) of detectable HBs Ag,
  * Chronic hepatitis B with serological remission HbsAg-negative , HB DNA-negative,
  * With or without association with acute or chronic hepatitis D.
* HCV-positive patients

  * Chronic hepatitis C defined by the positivity for anti-HCV antibodies for at least 6 months and positive HCV-RNA
  * Acute hepatitis C defined by the recent appearance of HCV RNA (less than 6 months) in patients with risk factors (with or without positive antibodies)
  * Patients with cured hepatitis C defined by long-term eradication, either spontaneous, a positive anti-HCV antibodies associated to a negative RNA at two collection - 6 months interval time; either treatment defined by negative viremia 3 month after end of treatment.

Exclusion Criteria:

* HIV co-infected patients are not eligible to the cohort.
* So-called vulnerable populations (minors, people under guardianship or protection, or a private individual under protection from making legal or administrative decisions)
* Treatment ongoing hepatitis C during or stopped since less than 3 months
* Patients end of life
* Woman whose pregnancy is known

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBV-positive patients and/or HCV-positive patients
Sampling Method: Non-Probability Sample
Enrollment: 20902 (Actual)
Dates: Start 2012-08-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
There is no specific primary outcome measure but we indicated below (see Description) a list of potential outcome measures according to the objectives. | From recruitment to the end of the cohort, with a minimum of one medical visit per year (the duration of follow-up is 7-8 years)
  * Effectiveness of HCV or HBV treatments: Virological response, seroconversion, loss of agHbS, liver fibrosis or clinical response (including quality of life), safety.
  * Prognostic factors of HCV or HBV infection: liver fibrosis, cirrhosis, clinical or biological event.
  * Biomarker studies: Virological response, seroconversion, loss of agHbS, liver fibrosis, clinical or biological event, safety
  * Cost-effectiveness studies: cost perYLS, cost per QALY

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas POL, MD, PhD, Principal Investigator — Hôpital Cochin, PARIS
Locations (1):
- Multiple Locations, France

REFERENCES:
- [Derived] Lotto M, Ramier C, Carrat F, Perieres L, Delaroque-Astagneau E, Nicol J, Marcellin F, Zoulim F, Di Beo V, Bertheau M, Pol S, Protopopescu C, Bourliere M, Carrieri P; ANRS/AFEF CO22 HEPATHER Study Group. Mortality risk in migrant and non-migrant individuals with chronic hepatitis B virus infection: a French hospital-based cohort study (ANRS CO22 HEPATHER). BMC Glob Public Health. 2025 Jul 1;3(1):58. doi: 10.1186/s44263-025-00173-7. PMID 40598581
- [Derived] Barre T, Parlati L, Bourliere M, Ramier C, Marcellin F, Protopopescu C, Di Beo V, Moins C, Dorival C, Nicol J, Zucman-Rossi J, Mathurin P, Larrey D, Boursier J, Carrat F, Carrieri P; ANRS/AFEF Hepather Study group. Socioeconomic Deprivation Weighs Heavily on Liver Fibrosis and Mortality After Hepatitis C Cure (ANRS CO22 Hepather). J Viral Hepat. 2024 Dec;31(12):830-846. doi: 10.1111/jvh.14006. Epub 2024 Sep 10. PMID 39252600
- [Derived] Poynard T, Lacombe JM, Deckmyn O, Peta V, Akhavan S, Zoulim F, de Ledinghen V, Samuel D, Mathurin P, Ratziu V, Thabut D, Housset C, Fontaine H, Pol S, Carrat F. External Validation of LCR1-LCR2, a Multivariable Hepatocellular Carcinoma Risk Calculator, in a Multiethnic Cohort of Patients With Chronic Hepatitis B. Gastro Hep Adv. 2022 May 25;1(4):604-617. doi: 10.1016/j.gastha.2022.02.008. eCollection 2022. PMID 39132068
- [Derived] Barre T, Bourliere M, Parlati L, Ramier C, Marcellin F, Protopopescu C, Di Beo V, Cagnot C, Dorival C, Nicol J, Zoulim F, Carrat F, Carrieri P; ANRS/AFEF Hepather Study group. Hepatitis C virus cure from direct-acting antivirals and mortality: Are people with and without a history of injection drug use in the same boat? (ANRS CO22 Hepather cohort). Drug Alcohol Rev. 2024 Mar;43(3):718-731. doi: 10.1111/dar.13802. Epub 2023 Dec 22. PMID 38133601
- [Derived] Carrieri P, Bourliere M, Di Beo V, Lusivika-Nzinga C, Ramier C, Antwerpes S, Protopopescu C, Lacombe JM, Pol S, Fontaine H, Mourad A, Carrat F, Duracinsky M, Marcellin F; ANRS/AFEF HEPATHER Study Group. Impaired health-related quality of life in the HCV cure era: who is concerned? (ANRS CO22 HEPATHER French cohort). Qual Life Res. 2023 Dec;32(12):3427-3438. doi: 10.1007/s11136-023-03496-w. Epub 2023 Aug 16. PMID 37587323
- [Derived] Sotty J, Bablon P, Lekbaby B, Augustin J, Girier-Dufournier M, Langlois L, Dorival C, Carrat F, Pol S, Fontaine H, Sarica N, Neuveut C, Housset C, Kremdsorf D, Schnuriger A, Soussan P. Diversity of the nucleic acid forms of circulating HBV in chronically infected patients and its impact on viral cycle. Hepatol Int. 2022 Dec;16(6):1259-1272. doi: 10.1007/s12072-022-10389-6. Epub 2022 Aug 4. PMID 35927368
- [Derived] Barre T, Carrat F, Ramier C, Fontaine H, Di Beo V, Bureau M, Dorival C, Larrey D, Delarocque-Astagneau E, Mathurin P, Marcellin F, Petrov-Sanchez V, Cagnot C, Carrieri P, Pol S, Protopopescu C; ANRS/AFEF Hepather study group. Cannabis use as a factor of lower corpulence in hepatitis C-infected patients: results from the ANRS CO22 Hepather cohort. J Cannabis Res. 2022 Jun 11;4(1):31. doi: 10.1186/s42238-022-00138-9. PMID 35690798
- [Derived] Pageaux GP, Nzinga CL, Ganne N, Samuel D, Dorival C, Zoulim F, Cagnot C, Decaens T, Thabut D, Asselah T, Mathurin P, Habersetzer F, Bronowicki JP, Guyader D, Rosa I, Leroy V, Chazouilleres O, de Ledinghen V, Bourliere M, Causse X, Cales P, Metivier S, Loustaud-Ratti V, Riachi G, Alric L, Gelu-Simeon M, Minello A, Gournay J, Geist C, Tran A, Abergel A, Portal I, d'Alteroche L, Raffi F, Fontaine H, Carrat F, Pol S; French ANRS CO22 Hepather Cohort. Clinical outcomes after treatment with direct antiviral agents: beyond the virological response in patients with previous HCV-related decompensated cirrhosis. BMC Infect Dis. 2022 Jan 27;22(1):94. doi: 10.1186/s12879-022-07076-0. PMID 35086481
- [Derived] Poynard T, Lacombe JM, Deckmyn O, Peta V, Akhavan S, de Ledinghen V, Zoulim F, Samuel D, Mathurin P, Ratziu V, Thabut D, Housset C, Fontaine H, Pol S, Carrat F. External validation of LCR1-LCR2, a multivariable HCC risk calculator, in patients with chronic HCV. JHEP Rep. 2021 Apr 24;3(4):100298. doi: 10.1016/j.jhepr.2021.100298. eCollection 2021 Aug. PMID 34142073
- [Derived] Barre T, Ramier C, Di Beo V, Carrat F, Fontaine H, Marcellin F, Carrieri P, Pol S, Protopopescu C; ANRS/AFEF Hepather study group. Liver fibrosis and all-cause mortality in chronic HCV-infected diabetic patients: A paradoxical association? (ANRS CO22 HEPATHER). Liver Int. 2021 Jul;41(7):1694-1698. doi: 10.1111/liv.14949. Epub 2021 May 28. No abstract available. PMID 33993651
- [Derived] Chalouni M, Pol S, Sogni P, Fontaine H, Lacombe K, Marc-Lacombe J, Esterle L, Dorival C, Bourliere M, Bani-Sadr F, de Ledinghen V, Zucman D, Larrey D, Salmon D, Carrat F, Wittkop L; ANRS CO13 HEPAVIH and ANRS CO22 HEPATHER cohort study groups. Increased mortality in HIV/HCV-coinfected compared to HCV-monoinfected patients in the DAA era due to non-liver-related death. J Hepatol. 2021 Jan;74(1):37-47. doi: 10.1016/j.jhep.2020.08.008. Epub 2020 Aug 14. PMID 32798585
- [Derived] Laurain A, Metivier S, Haour G, Larrey D, Dorival C, Hezode C, Zoulim F, Marcellin P, Bourliere M, Zarski JP, Thabut D, Alric L, Ganne-Carrie N, Cales P, Bronowicki JP, Riachi G, Geist C, Causse X, Abergel A, Chazouilleres O, Mathurin P, Guyader D, Samuel D, Tran A, Loustaud-Ratti V, Petrov-Sanchez V, Diallo A, Luzivika-Nzinga C, Fontaine H, Carrat F, Pol S; ANRS/AFEF HEPATHER study group. Safety and efficacy of the combination simeprevir-sofosbuvir in HCV genotype 1- and 4-mono-infected patients from the French ANRS CO22 hepather cohort. BMC Infect Dis. 2019 Apr 2;19(1):300. doi: 10.1186/s12879-019-3923-5. PMID 30940090
- [Derived] Carrat F, Fontaine H, Dorival C, Simony M, Diallo A, Hezode C, De Ledinghen V, Larrey D, Haour G, Bronowicki JP, Zoulim F, Asselah T, Marcellin P, Thabut D, Leroy V, Tran A, Habersetzer F, Samuel D, Guyader D, Chazouilleres O, Mathurin P, Metivier S, Alric L, Riachi G, Gournay J, Abergel A, Cales P, Ganne N, Loustaud-Ratti V, D'Alteroche L, Causse X, Geist C, Minello A, Rosa I, Gelu-Simeon M, Portal I, Raffi F, Bourliere M, Pol S; French ANRS CO22 Hepather cohort. Clinical outcomes in patients with chronic hepatitis C after direct-acting antiviral treatment: a prospective cohort study. Lancet. 2019 Apr 6;393(10179):1453-1464. doi: 10.1016/S0140-6736(18)32111-1. Epub 2019 Feb 11. PMID 30765123
- [Derived] Pol S, Bourliere M, Lucier S, Hezode C, Dorival C, Larrey D, Bronowicki JP, Ledinghen VD, Zoulim F, Tran A, Metivier S, Zarski JP, Samuel D, Guyader D, Marcellin P, Minello A, Alric L, Thabut D, Chazouilleres O, Riachi G, Bourcier V, Mathurin P, Loustaud-Ratti V, D'Alteroche L, Fouchard-Hubert I, Habersetzer F, Causse X, Geist C, Rosa I, Gournay J, Saillard E, Billaud E, Petrov-Sanchez V, Diallo A, Fontaine H, Carrat F; ANRS/AFEF HEPATHER study group. Safety and efficacy of daclatasvir-sofosbuvir in HCV genotype 1-mono-infected patients. J Hepatol. 2017 Jan;66(1):39-47. doi: 10.1016/j.jhep.2016.08.021. Epub 2016 Sep 10. PMID 27622858
- See also: Related Info — http://www.anrs.fr